CLINICAL TRIAL: NCT06541015
Title: TENS (Transcutaneous Electrical Nerve Stimulation): Effect of Transcutaneous Spinal Direct Current Stimulation on Lower Limb Reflex, Volitional, and Functional Movement Post-stroke
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation on Post-stroke Patients
Acronym: TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Yasin Dhaher, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2018-0431
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke; Anterior Circulation Stroke of Uncertain Pathology
Keywords: Single unilateral stroke with single lower limb hemiparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Post Stroke - individuals with history of single unilateral stroke (>6 months since onset) (Experimental): Individuals, aged 18-80, male or female, with a history of single unilateral stroke with subsequent lower limb hemiparesis on either side (>6 months since onset)
  Interventions: Device: InTENSity 10 TENS Stimulator

INTERVENTIONS:
Device: InTENSity 10 TENS Stimulator — InTENSity 10 TENS stimulator is a portable electrotherapy device featuring Transcutaneous Electrical Nerve Stimulation (TENS) therapeutic device. The stimulator sends a gentle electrical current to underlying nerves and muscle group via electrodes applied on the skin. The parameters of device are controlled by the buttons.

SUMMARY:
The subjects will be asked to attend minimum 15 separate sessions, 6 for testing changes in reflex behaviors, 3 for testing changes in the influence of descending motor tracts on spinal motor neurons, 3 for each testing functional movement in response to a trip event and cross-tilt walking adaptation pattern, as part of their participation in the research study. The estimated amount of time to enroll and collect the data for each of the subjects is four months' time. The data will be analyzed and ready for grant preparation (if successful) in approximately four months after the start of the study.

DETAILED DESCRIPTION:
The subjects will be asked to attend minimum 15 separate sessions, 6 for testing changes in reflex behaviors, 3 for testing changes in the influence of descending motor tracts on spinal motor neurons, 3 for each testing functional movement in response to a trip event and cross-tilt walking adaptation pattern, as part of their participation in the research study. During the first session, the subjects will be screened and informed about the research study, so they can consent to their participation. They will also be oriented to the lab, the equipment, as well as the research team. Following the orientation, the remaining time will consist of approximately 3 hours of data collection. The remaining will last approximately 3 hours and consist of the completion of data collection. Additional sessions after 15 sessions will be optional and will be reserved for completing data collection if the subject is unable to complete a trial session or to analyze for test retest variability within the subject population. The estimated amount of time to enroll and collect the data for each of the subjects is four months' time. The data will be analyzed and ready for grant preparation (if successful) in approximately four months after the start of the study.

ELIGIBILITY:
Post Stroke Cohort:

Inclusion Criteria:

* History of single unilateral stroke with subsequent lower limb hemiparesis on either side (> 6 months since onset)
* Ability to walk as part of activities of daily living
* Age between 18 and 80

Exclusion Criteria:

* Presence of concurrent severe medical illness including unhealed pressure sore, active or untreated infection, thromboembolic disease, severe contracture, osteoporosis, heterotropic classification, lower limb fracture, severe pulmonary disease or cardiovascular instability, uncontrolled seizure, uncontrolled diabetes
* History of any neurological injury other than a single stroke
* Has received a Botox injection in the lower extremity within the last 4 months
* Any cognitive deficit that would prevent informed consent or ability to perform the experiment
* History of prior injury or surgery to the hip or knee
* Presence of significant lower extremity edema - Presence of cardiac pacemaker or any other electrically implanted device - Use of braces limiting harness/Lokomat fit (Any spinal orthoses such as TLSO, HALO)
* Weight greater than 300 pounds
* Adults unable to consent, infants, children, teenagers, pregnant women and prisoners will not be included in the study
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse
* Actively taking medications with agents known to increase (e.g. amphetamines) or decrease motor system excitability
* Suffered a concussion in the last 6 months.
* Unexplained headaches

Healthy Cohort:

Inclusion Criteria:

* No history of stroke, cerebral palsy, injury or surgery to the lower limb.
* Currently not taking any central nervous system (CNS) affecting medication.
* Ability to walk as part of activities of daily living
* Age between 18 and 80

Exclusion Criteria:

* Presence of concurrent severe medical illness including unhealed pressure sore, active or untreated infection, thromboembolic disease, severe contracture, osteoporosis, heterotropic classification, lower limb fracture, severe pulmonary disease or cardiovascular instability, uncontrolled seizure, uncontrolled diabetes
* History of any neurological injury
* Taking any medication affecting change in CNS
* Any cognitive deficit that would prevent informed consent or ability to perform the experiment
* History of prior injury or surgery to the hip or knee
* Presence of significant lower extremity edema - Presence of cardiac pacemaker or any other electrically implanted device - Use of braces limiting harness/Lokomat fit (Any spinal orthoses such as TLSO, HALO)
* Weight greater than 300 pounds
* Adults unable to consent, infants, children, teenagers, pregnant women and prisoners will not be included in the study
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse
* Actively taking medications with agents known to increase (e.g. amphetamines) or decrease motor system excitability
* Suffered a concussion in the last 6 months.
* Unexplained headaches
* Has received a Botox injection in the lower extremity within the last 4 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflex Testing | 3 months
  Test if tsDCS (transcutaneous spinal direct current stimulation) has any beneficial effect on reflexes in post-stroke individuals
Walking Testing | 3 months
  Test if tsDCS (transcutaneous spinal direct current stimulation) has any beneficial effect on walking in post-stroke individuals
Adaptation Testing | 3 months
  Test if tsDCS (transcutaneous spinal direct current stimulation) has any beneficial effect on adaptation pattern in post-stroke individuals

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Dhaher, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No